CLINICAL TRIAL: NCT01351090
Title: A Phase 2, Double-blind, Randomized Study of the Safety, Tolerability and Analgesic Efficacy of Multiple Doses of Ketorolac Tromethamine Administered Intranasally for Postoperative Pain
Brief Title: Study of the Safety, Tolerability and Analgesic Efficacy of Multiple Doses of Ketorolac Tromethamine (IN) for Postoperative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: David Bregman, M.D., Ph.D., Luitpold Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROX 2001-03
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ketorolac tromethamine (5%) (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Ketorolac tromethamine (15%) (Experimental)
  Interventions: Drug: Ketorolac tromethamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac tromethamine — 10 mg Intranasal (2 x 100 uL of a 5% solution)
  Arms: Ketorolac tromethamine (5%)
Drug: Ketorolac tromethamine — 30 mg Intranasal (2 x 100 uL of a 15% solution)
  Arms: Ketorolac tromethamine (15%)
Drug: Placebo — Intranasal
  Arms: Placebo

SUMMARY:
This was a randomized, double blind, placebo-controlled study in subjects who have undergone major surgery. Each subject's study participation consisted of a screening visit, a 2-day treatment period, and a follow-up visit. Following surgery, subjects were randomly assigned to receive intranasally (IN) ketorolac 10 mg, IN ketorolac 30 mg, or placebo when the pain intensity (PI) rating equaled at least 40 on a 100-mm visual analog scale (VAS). Thereafter, subjects received study drug every 8 hours, with the last dose given at 40 hours. For pain not relieved by the study drug, the subjects had access to morphine sulfate (MS) administered via patient controlled analgesia (PCA).

The primary objective was to evaluate the analgesic efficacy of multiple intranasal (IN) doses of ketorolac over 2 days. The secondary objective was to evaluate the safety and tolerability of this dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 years or older
* Body weight > or = 100 pounds (45.4 kg) and < or = 300 pounds (136.1 kg)
* Women of childbearing potential must have had a negative serum pregnancy test result prior to entry into the study
* Able to provide written informed consent
* At least moderate pain as determined by a PI score of > or = 40 mm on a 100-mm VAS
* Expected to remain in the hospital for at least 48 hours
* Willing and able to comply with all testing and requirements defined in the protocol
* Willing and able to complete the posttreatment visit

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or ethylene diamine tetraacetic acid (EDTA)
* Allergic reaction to aspirin or other nonsteroidal anti-inflammatory drug (NSAIDs)
* Current upper respiratory tract infection or other respiratory tract condition that could interfere with the absorption of the nasal spray or with the assessment of adverse events
* Use of any IN product within 24 hours prior to study entry
* Clinically significant abnormality on screening laboratory tests
* History of cocaine use resulting in nasal mucosal damage
* Active peptic ulcer disease, recent (defined as within 6 months) gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Advanced renal impairment or a risk for renal failure due to volume depletion
* A history of any other clinically significant medical problem, which in the opinion of the investigator would interfere with study participation
* Participation within 30 days of study entry or within 5 times the half-life, whichever is longer, in another investigational drug study
* Allergy or significant reaction to opioids
* Pregnancy or breastfeeding
* Previous participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Chair — ICON Development Solutions
Locations (1):
- Waikato Clinical Research, Hamilton, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period - October 2001 through August 2002 Locations - Hospitals
Pre-assignment Details: Subjects must have been requesting pain medication and have at lease moderate pain defined as a score of at least 40 mm on a 100-mm VAS.
Groups:
- Ketorolac IN 10 mg: 10 mg Intranasal (2 x 100 uL of a 5% solution)
- Ketorolac IN 30 mg: 30 mg Intranasal (2 x 100 uL of a 15% solution)
- Placebo Vehicle IN: Intranasal placebo
Period: Overall Study
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Started | 43 | 42 | 42
Completed | 32 | 31 | 36
Not Completed | 11 | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN | Total
Number analyzed (Participants) | 43 | 42 | 42 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 29 | 25 | 91
  >=65 years | 6 | 13 | 17 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 49.7 (2.1) | 52.8 (2.5) | 56.7 (2.5) | 53.0 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 24 | 85
  Male | 11 | 13 | 18 | 42
Region of Enrollment [Number; unit: participants]
  New Zealand | 43 | 42 | 42 | 127

OUTCOME MEASURES:

1. Primary Outcome: Total Morphine Sulfate (MS) Use in Milligrams by Patient-controlled Analgesia (PCA) Through 24 Hours
Time Frame: 8-hour intervals from the start of dosing through 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Number analyzed (Participants) | 41 | 41 | 41
mg | 54.32 (6.36) | 37.77 (4.98) | 56.45 (4.82)

2. Secondary Outcome: Total MS Use in Milligrams by PCA From the Start of Dosing Through 48 Hours
Time Frame: 8-hour intervals from the start of dosing through 48 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Number analyzed (Participants) | 38 | 35 | 39
mg | 78.66 (11.20) | 61.39 (10.79) | 87.87 (9.36)

3. Secondary Outcome: Total MS Use in Milligrams by PCA From 24 Hours After the Start of Dosing Through 48 Hours
Time Frame: 8-hour intervals from 24 hours after the start of dosing through 48 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Number analyzed (Participants) | 38 | 35 | 39
mg | 28.25 (5.67) | 23.11 (5.31) | 32.61 (4.77)

4. Secondary Outcome: Pain Intensity Difference (PID) Scores
Description: Ratings of Pain Intensity (PI) were made using a 100-mm Visual Analog Scale (VAS) on which 0 = no pain and 100 = worst pain possible. PID was calculated by subtracting the posttreatment score from the baseline score, where the baseline score was the PI rating made prior to the first dose of study medication.
Time Frame: 6 hours after study drug administration
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Number analyzed (Participants) | 43 | 42 | 42
units on a scale | 34.1 (2.7) | 38.9 (2.1) | 29.1 (2.3)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Ketorolac IN 10 mg | Ketorolac IN 30 mg | Placebo Vehicle IN
Serious Adverse Events (participants affected / at risk) | 3/43 | 5/42 | 1/42
Other Adverse Events (participants affected / at risk) | 43/43 | 39/42 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac IN 10 mg (N=43) | Ketorolac IN 30 mg (N=42) | Placebo Vehicle IN (N=42)
Pulmonary embolism (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombus in popliteal vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ketorolac IN 10 mg (N=43) | Ketorolac IN 30 mg (N=42) | Placebo Vehicle IN (N=42)
Anemia NOS (Blood and lymphatic system disorders) | 12 | 11 | 14
Tachycardia NOS (Cardiac disorders) | 7 | 8 | 17
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 8 | 11 | 10
Dyspesia (Gastrointestinal disorders) | 3 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 25 | 19 | 20
Vomiting NOS (Gastrointestinal disorders) | 12 | 12 | 11
Pyrexia (General disorders) | 24 | 14 | 26
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Dizziness (Nervous system disorders) | 7 | 6 | 5
Headache (Nervous system disorders) | 15 | 9 | 9
Somnolence (Nervous system disorders) | 9 | 1 | 5
Urinary retention (Renal and urinary disorders) | 1 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 5
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 8 | 4 | 10
Hypotension NOS (Vascular disorders) | 4 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No